CLINICAL TRIAL: NCT04759365
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 1 Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Study of Oral ASN51 in Healthy Young Adult and Elderly Subjects and Elderly Subjects With Alzheimer's Disease
Brief Title: Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Study of Oral ASN51 in Healthy Subjects and Subjects With Alzheimer's Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Delays with sites, identifying/enrolling patients, impact of COVID, staffing, and duration
Sponsor: Asceneuron Pty Ltd. (Industry)
Collaborators: Asceneuron S.A. (Industry); Neuroscience Trials Australia (Other)
Responsible Party: Sponsor
Organization: Asceneuron S.A. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASN51-101
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASN51 (Experimental): ASN51 will be administered as an oral capsule
  Interventions: Drug: ASN51
- Placebo (Placebo Comparator): Placebo will be administered as an oral capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASN51 — ASN51 formulation for oral capsule
  Arms: ASN51
Drug: Placebo — Placebo formulation for oral capsule
  Arms: Placebo

SUMMARY:
ASN51-101 is a randomized, double-blind, placebo-controlled, phase 1 first in human (FIH) safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) study of oral ASN51 in healthy young adult and elderly subjects and elderly subjects with AD. The study is comprised of three parts (Part 1, Part 2, and Part 3).

DETAILED DESCRIPTION:
Part 1:

Five (5) single-ascending oral doses will be administered to 40 healthy adult male or female subjects (aged 18-55 years, inclusive). Escalation to the next higher dose level may occur only after evaluation of the safety and PK results of the previous dose level (at least 6 evaluable subjects). Within each cohort, 6 subjects will receive one dose of ASN51, and 2 subjects will receive one dose of matching placebo. Based on this interim safety evaluation, dose levels may be revised.

Part 2:

Multiple ascending oral doses will be administered to 24 healthy elderly subjects (aged 55 - 80 years, inclusive) in 3 sequential dosing groups (8 subjects in each dosing group). Six (6) subjects will receive ASN51 and two (2) subjects will receive matching placebo in each dosing group (cohort) for 10 days. Escalation to the next higher dose level may occur only after evaluation of the safety and PK results of the previous dose level (at least 6 evaluable subjects). Based on this interim safety evaluation, dose levels may be revised.

Treatment of the subjects of each cohort will be administered as follows:

Day 1 - 9: Twice daily (BID) dosing (or once daily (QD) dosing); to be defined after Part 1 (SAD) of ASN51 or placebo.

Day 10: Only one dose will be administered in the morning of Day 10 Selection of the dosing regimen and dose levels to be administered in Part 2 will be made by the safety review committee (SRC), depending on the results of Part 1.

Part 3:

Multiple oral doses will be administered to 12 AD subjects (aged 55-85, inclusive) in a single dosing group for 10 days. Eight (8) AD subjects will receive ASN51 and four (4) AD subjects will receive placebo in that dosing group (cohort). Selection of the dose level to be administered in Part 3 will be made by the SRC and will depend on the results of study Part 1 (SAD) and Part 2 (MAD), and will be below the maximum tolerated dose administered to healthy subjects in Part 2.

Treatment of the AD subjects will be administered as follows:

Day 1 - 9: Twice daily (BID) dosing (or once daily (QD) dosing); to be defined after Part 2 (MAD) of ASN51 or placebo.

Day 10: Only one dose will be administered in the morning of Day 10. Selection of the dosing regimen and dose level to be administered in Part 3 will be made by the safety review committee (SRC), depending on the results of both Part 1 and Part 2.

ELIGIBILITY:
Part 1 and Part 2 Only:

Inclusion Criteria:

1. Healthy as determined by the Investigator, based on a medical evaluation including medical history, physical examination, neurological examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if, in the opinion of the Investigator, the finding is (a) unlikely to introduce additional risk to the subject, (b) will not interfere with study procedures or confound study results, and (c) is not otherwise exclusionary (see Exclusion Criteria).
2. Men and women aged 18-55 years, inclusive, at Screening (Part 1) or 55-80 years, inclusive, at Screening (Part 2)
3. Subject must understand the nature of the study and provide signed and dated written informed consent in accordance with local regulations before the conduct of any study-related procedures.
4. Able to complete all study related testing and evaluations
5. Women (Part 1 only) and men of child-bearing potential with partners of child-bearing potential must agree to use highly effective contraception. Contraception should consist of: (1) a condom for the male participant or partner of a female participant, combined with (2) a highly effective method of contraception (e.g., a hormonal method associated with suppression of ovulation, an intrauterine device [IUD]) for the female participant or partner of a male participant. Abstinence from heterosexual intercourse should only be used in place of contraception when this is consistent with the usual and preferred lifestyle of the participant. For male subjects, contraception should continue for 90 days after the last dose of investigational medicinal product (IMP, one spermatic cycle). Male subjects should agree to refrain from sperm donation throughout this same period.
6. Women of non-childbearing potential must be post-menopausal (the last menstrual period was at least 12 months ago, and follicle-stimulating hormone [FSH] at Screening confirms post-menopausal status), or have no uterus, ovaries, or fallopian tubes (or have their fallopian tubes tied). All women must have a negative pregnancy test result before administration of test article. Women who are surgically sterile must provide documentation of the procedure by an operative report or by ultrasound.
7. Body weight > 50.0 kg for men and > 50 kg for women and Body Mass Index (BMI) within the range 18.5-30.0 kg/m2, inclusive.
8. Subject must be, in the opinion of the Investigator, able to participate in all scheduled evaluations, likely to complete all required tests, and likely to be compliant.
9. Subjects is fluent in the local language.
10. Subject agrees not to post any personal medical data related to the study or information related to the study on any website or social media site (e.g., Facebook, Twitter, etc.) until the trial has been completed, this does not include information about participating in a clinical study in general.
11. [Part 2 only] Subject is able to undergo Lumbar Puncture (LP)

Exclusion Criteria:

1. A positive urine drug screen/alcohol breath test at Screening or Day -1.
2. Any history of intellectual disability or psychiatric disorders, including substance use disorders, according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria, except a history of mild depression/anxiety that has been resolved for at least the past 12 months.
3. A positive Hepatitis B surface antigen, Hepatitis C antibody, or Human Immunodeficiency Virus (HIV) antibody test at Screening.
4. Alanine aminotransferase or aspartate aminotransferase levels greater than 1.5 times the upper limit of normal (ULN) at Screening or between Screening and first dose administration.
5. Frequent use of any tobacco-containing (e.g., cigar, cigarette, or snuff) or nicotine-containing product (e.g., nicotine chewing gum, nicotine plasters, or other product used for smoking cessation) within 3 months prior to 1 week before study drug administration. Frequent use is defined as more than 10 cigarettes or equivalent per week. Use of any tobacco or nicotine-containing product is prohibited from 1 week prior to study drug administration throughout the study (final visit).
6. History of regular alcohol consumption within the last 12 months, defined as an average weekly intake of >21 alcoholic drinks/week for men or >14 alcoholic drinks/week for women.
7. Regularly consumed (e.g., more days than not) excessive quantities of xanthine-containing beverages (e.g., more than five cups of coffee or the equivalent per day) within 30 days prior to Day -1.
8. Received or used an investigational product (including placebo) or device within the following time period prior to Day -1 in the current study: 90 days, 5 half-lives, or twice the duration of the biological effect of the investigational product (whichever is longer).
9. Use of prescription or non-prescription drugs, vitamins, herbal, and dietary supplements (including St John's Wort) within 7 days (or 28 days if the drug is a potential hepatic enzyme inducer) or 5 half-lives (whichever is longer) prior to Day -1.
10. History of clinically significant sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates their participation.
11. Loss of more than 400 mL of blood within 3 months prior to Day -1, i.e., blood donor
12. A positive serum pregnancy test or lactation.
13. Hearing test result considered unacceptable for auditory ERP P300 assessment.
14. A history or presence of any disease, condition, or surgery likely to affect drug absorption, distribution, metabolism, or excretion. Subjects with a history of cholecystectomy should be excluded.
15. A history or presence of a clinically significant hepatic, renal, gastrointestinal, cardiovascular, endocrine, pulmonary, ophthalmologic, immunologic, hematologic, dermatologic, or neurologic abnormality.
16. A clinically significant abnormality on physical examination, neurological examination, electrocardiogram (ECG), or laboratory evaluations at Screening or between Screening and first dose administration.
17. A corrected QT interval measurement corrected according to the Fridericia rule (QTcF) > 450 msec during controlled rest at screening or between screening and first dose administration, or family history of long QT syndrome.
18. Any clinically significant abnormalities in rhythm, conduction, or morphology of the resting ECG and any abnormalities in the 12-lead ECG that, in the judgement of the Investigator or Medical Monitor, may interfere with the interpretation of QTc interval changes, including abnormal ST-T-wave morphology or left ventricular hypertrophy.
19. PR (PQ) interval shortening < 120 msec (PR < 120 msec but > 110 msec is acceptable if there is no evidence of ventricular pre-excitation).
20. PR (PQ) interval prolongation (> 220 msec), intermittent second- (Wenckebach block while asleep or in deep rest is not exclusionary) or third-degree AV block.
21. Persistent or intermittent complete bundle branch block (BBB), incomplete bundle branch block (IBBB), or intraventricular conduction delay (IVCD) with QRS > 120 msec.
22. A clinically significant vital signs abnormality at Screening or Day -1 This includes, but is not limited to, the following, in the sitting position (3 measurements, each 5 minutes apart): (a) systolic blood pressure < 90 or >140 mmHg, (b) diastolic blood pressure < 50 or > 95 mmHg, or (c) heart rate < 45 or > 100 beats per minute.
23. Significant (> 10%) weight loss or gain within 30 days prior to Day -1
24. A history of seizure.
25. A history of head trauma, with loss of consciousness, except for minor head trauma that occurred at least 20 years prior to first dose.
26. A history of symptomatic orthostatic hypotension (i.e., postural syncope) or symptomatic orthostatic hypotension at Screening.
27. A history of neuroleptic malignant syndrome.
28. A history of chronic urinary tract infections.
29. The subject is, in the opinion of the Investigator or Medical Monitor, unlikely to comply with the protocol or is unsuitable for any reason, e.g., known issues with ability to swallow size 00 capsules.
30. Currently employed by Asceneuron SA or by a clinical trial site participating in this study, or a first-degree relative of an Asceneuron SA employee or of an employee at a participating clinical trial site.
31. Unsatisfactory venous access.
32. Identification of suicide risk in the Columbia-Suicide Severity Rating Scale (C-SSRS).
33. Part 2 only: Abnormal exercise ECG in relation to age.

Part 3 Only:

Inclusion Criteria

1. Between 55-85 years of age, inclusive.
2. Mild cognitive impairment due to AD or Mild-to-moderate AD dementia, Mini-Mental State Examination (MMSE) 14-27 and Clinical Dementia Rating (CDR) 0.5, 1 or 2 at the Screening Visit.
3. Clinical diagnosis of mild cognitive impairment or dementia, due probably to AD, by Revised National Institute on Aging-Alzheimer's Association criteria.
4. Reliable and capable support person/caregiver.
5. Able to undergo Lumbar Puncture (LP) and complete all study related testing and evaluations.
6. Women of non-childbearing potential must be post-menopausal [the last menstrual period was at least 12 months ago, and FSH at Screening confirms post-menopausal status], or have no uterus, ovaries, or fallopian tubes; or have their fallopian tubes tied. All women must have a negative pregnancy test result before administration of test article. Women who are surgically sterile must provide documentation of the procedure by an operative report or by ultrasound.
7. Women and men of child-bearing potential with partners of child-bearing potential must agree to use highly effective contraception. Contraception should consist of: (1) a condom for the male participant or partner of a female participant, combined with (2) a highly effective method of contraception (e.g., a hormonal method associated with suppression of ovulation, an IUD) for the female participant or partner of a male participant. Abstinence from heterosexual intercourse should only be used in place of contraception when this is consistent with the usual and preferred lifestyle of the participant. For male subjects, contraception should continue for 90 days after the last dose of IMP (one spermatic cycle). Male subjects should agree to refrain from sperm donation throughout this same period.
8. Treatment-free or receiving stable acetylcholinesterase inhibitor (AChEI) treatment, defined as:

   * Subjects who are taking an approved AChEI for at least 2 weeks prior to the first Screening biomarker for efficacy assessment at a dose that is not anticipated to change through the study follow-up period, OR
   * Subjects who received an AChEI in the past and discontinued, e.g., due to tolerability issues, at least 5 half-lives or 30 days before the first Screening biomarker or efficacy assessment, whichever is longer.

Exclusion Criteria:

1. Receipt of any investigational drug or device within 8 weeks or 4 half-lives, whichever is longer, prior to randomization.
2. History of cardiovascular disease or at risk of stroke or heart attack, peripheral vascular intervention, atrial fibrillation, clinically relevant cardiac arrhythmias, or uncontrolled hypertension.
3. History within 2 years of Screening, or current diagnosis of the any of the following psychiatric disorders: Schizophrenia, schizoaffective disorder, bipolar disorder I, or alcohol abuse or dependence per DSM-5 criteria.
4. History of unexplained loss of consciousness, and seizures (excluding infant febrile seizures)
5. Ongoing infectious, metabolic, or systemic diseases affecting the central nervous system (CNS) (e.g. syphilis, untreated hypothyroidism, current vitamin B12 or folate deficiency, potentially clinically significant serum electrolyte disturbances, unstable diabetes mellitus (HbA1c > 10.5%); or other similar conditions.
6. History within 2 years of Screening, or current diagnosis of a chronic inflammatory disease (i.e., rheumatoid arthritis, systemic lupus, erythematosus, Crohn's disease, etc.).
7. A positive Hepatitis B surface antigen, Hepatitis C antibody, or Human Immunodeficiency Virus (HIV) antibody test at Screening.
8. The subject has received active amyloid or tau immunization at any time, or passive immunization within 12 months of Screening.
9. Intake of any of the prohibited medications listed below within the past 30 days or 5 half-lives, whichever is longer. Subjects need to stay off the medication during the trial.

   * For memantine, a 1-month drug-free period is required between the last dose received and Screening
   * Anticonvulsants
   * Neuroleptics (quetiapine and clozapine are allowed)
   * Centrally active anti-hypertensive drugs (e.g., clonidine, alpha-methyldopa, guanidine, or guanfacine)
   * Immunosuppressants or systemic corticosteroids >10 mg/day prednisone or equivalent
   * Anticoagulants

9. History or presence of brain MRI scans indicative of a neurologic disease other than AD or any other significant abnormality.

10. Subject has an atypical variant presentation of AD, if known from medical history, particularly non-amnestic AD.

11. History of treatment for cancer within the past 2 years. Subjects who have undergone curative excision of basal cell carcinoma or squamous cell carcinoma of the skin within the past 2 years are permitted.

12. Blood pressure and ECG parameters at Screening:

* Seated systolic blood pressure < 90 mmHg or > 150 mmHg; or diastolic blood pressure < 50 mmHg or > 95 mmHg
* ECG abnormalities on the screening ECG including: clinically significant conduction abnormalities, ischemic changes (e.g., prior Q-wave myocardial infarction and/or marked ischemic ST- and T-wave), arrhythmias (e.g., persistent or paroxysmal ventricular or supraventricular arrhythmias, including atrial fibrillation), or other ECG abnormalities that would pose unnecessary risk in the opinion of the Investigator
* QTc interval > 450 in males or > 470 in females utilizing Fredericia's correction (QTcF)

  13. Abnormal stress ECG in relation to age at Screening.

  14. Renal insufficiency (serum creatinine >177 μmol/L).

  15. Hepatic impairment with alanine aminotransferase or aspartate aminotransferase > 1.5 times the upper limit of normal, or Child-Pugh class B or C.

  16. Hearing test result considered unacceptable for auditory ERP P300 assessment.

  17. Positive urine or serum pregnancy test, lactating, or plans to become pregnant during the trial.

  18. Significant suicide risk as assessed by C-SSRS.

  19. Any condition that in the judgement of the Investigator would interfere with the ability to complete the trial, pose significant risk to subject safety, or potentially confound interpretation of trial results, e.g., known issues with ability to swallow size 5 capsules.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Up to 38 days

SECONDARY OUTCOMES:
PK parameter: The area under the concentration-time curve from time zero to time t of the last measured concentration above the limit of quantification (AUC0-t) in plasma | Up to 10 days
PK parameter: The area under the concentration-time curve from zero to infinity (AUC0-inf) in plasma | Up to 10 days
PK parameter: The maximum concentration (Cmax) at steady state in plasma | Up to 10 days
PK parameter: The time to reach maximum concentration (tmax) in plasma | Up to 10 days
PK parameter: The terminal elimination rate constant (λZ) with the respective half-life (t½) in plasma | Up to 10 days
PK parameter: The percentage of the extrapolated AUC in plasma | Up to 10 days
PK parameter: Area under the concentration-time curve from time zero to the end of the dosing interval (AUCtau) in plasma (Part 2 Day 1 only) | Up to 1 day
PK parameter: The minimal observed trough concentration (Cmin) at steady state in plasma | Up to 10 days
PK parameter: The average concentration (Cavg) at steady state in plasma | Up to 10 days
PK parameter: Accumulation Ratio: AUCtau at Day 10/ AUCtau at Day 1 in plasma | Up to 10 days
PK parameter: The mean cumulative amounts excreted (both in % of the administered dose and in mg ASN51) will be calculated both for Fe(0-72h) and Fe(0-tau) and Ae(0-72h) and Ae(0-tau), respectively | Up to 10 days
PK parameter: The area under the plasma concentration-time curve from time zero to time t of the last measured concentration above the limit of quantification (AUC0-t) in cerebrospinal fluid (CSF) | Up to 10 days
PK parameter: The area under the plasma concentration-time curve from zero to infinity (AUC0-∞) in CSF | Up to 10 days
PK Parameter: The maximum plasma concentration (Cmax) in CSF | Up to 10 days
PK parameter: The time to reach maximum plasma concentration (tmax) in CSF | Up to 10 days
PK parameter: The terminal elimination rate constant (λZ) with the respective half-life (t½) in CSF | Up to 10 days
PK parameter: The percentage of the extrapolated AUC in CSF | Up to 10 days
PK parameter: Area under the concentration-time curve from time zero to the end of the dosing interval (AUCtau) in CSF | Up to 10 days
PD parameter: Change from baseline in total and phosphorylated CSF tau | Up to 10 days
PD parameter: Change from baseline in quantitative electroencephalography power and the P300 event related potential (ERP) | Up to 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No